CLINICAL TRIAL: NCT01536613
Title: NovoMix® 30 FlexPen, Post Marketing Surveillance Study
Brief Title: Post Marketing Surveillance Study of Biphasic Insulin Aspart 30
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1883
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIAsp 30 users
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — The insulin dose and regimen were individualised at the physician's discretion. Insulin was administered by subcutaneous injection using an injection device

SUMMARY:
This study is conducted in Asia. The aim of this study is to review the safety and efficacy of biphasic insulin aspart 30 in post-marketing use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diabetes who did not have indications that are contraindicated in the product insert

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with diabetes who did not have indications that are contraindicated in the product insert
Sampling Method: Non-Probability Sample
Enrollment: 5346 (Actual)
Dates: Start 2004-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Change in body weight

SECONDARY OUTCOMES:
Change in fasting plasma glucose (FPG)
Change in HbA1c (glycosylated haemoglobin)
Occurrence of adverse events (non-serious and serious)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Seoul, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com